CLINICAL TRIAL: NCT01437241
Title: Virological Efficacy and Safety of Etravirine Plus 2 Active Nucleos(t)Ide Reverse-transcriptase Inhibitors (NRTIs) in HIV-1-infected Patients
Brief Title: Etravirine Plus 2 Analogs in HIV-infected Patients
Status: Completed | Type: Observational
Sponsor: Hospitales Universitarios Virgen del Rocío (Other)
Responsible Party: Principal Investigator, Luis F. Lopez-Cortes, M.d., Ph.D., Hospitales Universitarios Virgen del Rocío
Other Study IDs: LFL-ETR-2010-01
Record Dates: First submitted 2011-09-17; First posted 2011-09-20 (Estimated); Last update posted 2011-11-01 (Estimated); Status verified 2011-10

CONDITIONS: HIV-1-infection
Keywords: HIV-infection; Etravirine; Treatment; Non-nucleoside reverse-transcriptase inhibitor
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- etravirine: Antiretroviral regimens based on etravirine plus 2 active nucleos(t)ide reverse-transcriptase inhibitors (NRTIs)

SUMMARY:
The purpose of this study is to evaluate the virological and clinical efficacy of etravirine plus 2 active nucleos(t)ide reverse-transcriptase inhibitors (NRTIs) in HIV-infected patients. Additionally, the safety of these regimens, specially lipid profiles, will be assessed.

DETAILED DESCRIPTION:
Methods: prospective, single arm multicenter clinical trial without entry restrictions on plasma HIV-RNA (VL) or CD4 with a planned duration of 52 weeks.

The primary clinical endpoint is the percentage of subjects with therapeutic success on etravirine 400 mg/day (200 mg bid or 400 mg qd) plus 2 active NRTIs after 12 months. Efficacy data will be analyzed by on-treatment and by intention-to-treat analyses (noncomplete/missing equals failure), considering treatment failure as either treatment interruption whatever the reason (adverse events, death, or loss to follow-up) or virological failure, defined as inability to suppress the VL to less than 50 copies/ml after 24 weeks on treatment or a confirmed VL of more than 200 copies/ml in patients who had previously achieved a viral suppression or had an undetectable viral load at inclusion.

Patients missing two consecutive scheduled visits were considered lost to follow-up. The safety and tolerability of the studied medications will be evaluated by means of clinical adverse events, physical examination and laboratory results.

NRTIs prescribed as part of HAART were selected by the responsible physicians on the basis of previous antiretroviral treatments and/or genotypic resistance testing.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years, starting an antiretroviral regimen based on etravirine plus 2 NRTIs between January 2009 and June 2010, evidence of activity of all drugs on the basis of treatment history and genotypic resistance testing, informed consent, and at least one follow-up visit.

Exclusion Criteria:

* Genotypic resistance tests with evidence of resistance to any drug used, and concomitant use of drugs with potentially adverse interactions with etravirine pharmacokinetics, such as rifampin.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-infected patients who strated an antirretroviral regimen based on etravirine plus 2 NRTIs between January 2009 and June 2010
Sampling Method: Non-Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2009-01; Primary Completion 2011-07 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Virological efficacy | 52 weeks
  Percentage of subjects with therapeutic success at month 12. Efficacy data will be analyzed by on-treatment and by intention-to-treat considering treatment failure as either treatment interruption whatever the reason (adverse events, death, or loss to follow-up) or virological failure, defined as inability to suppress the VL to <50 copies/ml after 24 weeks or a confirmed VL of >200 copies/ml in patients who had previously achieved a viral suppression or had an undetectable viral load at inclusion. Patients missing two consecutive scheduled visits were considered lost to follow-up.

SECONDARY OUTCOMES:
Safety | 52 weeks
  The safety and tolerability of the studied medications will be evaluated by means of clinical adverse events, physical examination and laboratory results.

CONTACTS AND LOCATIONS:
Overall Officials: Luis F Lopez-Cortes, MD, PhD., Principal Investigator — Hospitales Universitarios Virgen del Rocio; Francisco Tellez-Perez, MD, Principal Investigator — Hospital de la Linea de la Concepcion; Antonio Vergara-Campos, MD, PhD., Principal Investigator — Hospital Universitario de Puerto Real; Milagros Garcia-Lazaro, MD, Principal Investigator — Hospital Universitario Reina Sofia de Cordoba; Jose Hernandez-Quero, MD, PhD., Principal Investigator — Hospital Universitario San Cecilio; Juan Pascuau-Liaño, MD, PhD., Principal Investigator — University Hospital Virgen de las Nieves; Miguel A Lopez-Ruz, MD, PhD, Principal Investigator — University Hospital Virgen de las Nieves; Mohamed O Mohamed-Balghata, MD, Principal Investigator — Hospital Universitario Ciudad de Jaén; Dr.Javier de la Torre-Lima, MD, PhD, Principal Investigator — Hospital Costa del Sol; Manuel Marquez Solero, MD, Principal Investigator — Hospital Universitario Virgen de la Victoria; Marcial delgado, MD, Principal Investigator — Hospital Universitario Carlos Haya; Fernando Lozano-León, MD, PhD., Principal Investigator — Hospital Universitario de Valme
Locations (11):
- Spain (11):
  - Hospital La Linea de la Concepción, La Linea de La Concepción, Cadiz
  - Hospital Universitario Puerto Real, Puerto Real, Cadiz
  - Hospital Universitario Reina Sofía, Córdoba, Cordoba
  - Hospital Universitario San Cecilio, Granada, Granada
  - Hospital Universitario Virgen de las Nieves, Granada, Granada
  - Hospital Ciudad de Jaén, Jaén, Jaen
  - Hospital Costa del Sol, Marbella, Malaga
  - Hospital Universitario Carlos Haya, Málaga, Malaga
  - Hospital Universitario Virgen de la Victoria, Málaga, Malaga
  - Hospital Universitario Virgen del Rocio, Seville, Sevilla
  - Hospital Universitario Virgen de Valme, Seville, Sevilla

REFERENCES:
- [Derived] Lopez-Cortes LF, Viciana P, Giron-Gonzalez JA, Romero-Palacios A, Marquez-Solero M, Martinez-Perez MA, Lopez-Ruz MA, de la Torre-Lima J, Tellez-Perez F, Delgado-Fernandez M, Garcia-Lazaro M, Lozano F, Mohamed-Balghata MO; Sociedad Andaluza de Enfermedades Infecciosas. Clinical and virological efficacy of etravirine plus two active Nucleos(t)ide analogs in an heterogeneous HIV-infected population. PLoS One. 2014 May 16;9(5):e97262. doi: 10.1371/journal.pone.0097262. eCollection 2014. PMID 24836963